CLINICAL TRIAL: NCT01569022
Title: A Randomized Cross Over Trial of Two Treatments for OSA in Veterans With PTSD
Brief Title: A Randomized Cross Over Trial of Two Treatments for Sleep Apnea in Veterans With Post-Traumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-005-11F
Record Dates: First submitted 2012-03-20; First posted 2012-04-02 (Estimated); Results first posted 2017-11-08 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Obstructive Sleep Apnea
Keywords: post traumatic stress disorder; continuous positive airway pressure; oral appliance
MeSH Terms: conditions — Sleep Apnea, Obstructive; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- CPAP First, MAD (Active Comparator): CPAP treatment for sleep apnea
  CPAP: CPAP Treatment for 12 weeks MAD: MAD treatment for 12 weeks
  Interventions: Device: CPAP; Device: MAD
- MAD First, CPAP (Experimental): MAD treatment for sleep apnea
  MAD: MAD Treatment for 12 weeks CPAP: CPAP treatment for 12 weeks
  Interventions: Device: CPAP; Device: MAD

INTERVENTIONS:
Device: CPAP — CPAP Treatment for 12 weeks
Device: MAD — MAD Treatment for 12 weeks

SUMMARY:
Sleep disturbances are cardinal features of Veterans with post traumatic stress disorder (PTSD). In particular, obstructive sleep apnea is reported to occur more frequently in patients with PTSD compared to those without PTSD and contribute to worsening cognitive and behavioral functions. Continuous positive airway pressure (CPAP) is considered the treatment of choice for OSA but adherence to CPAP in Veterans with PTSD is poor compared to the general population. The proposed study aims at comparing the efficacy, tolerability, and adherence of oral appliances-an alternative therapy to OSA- to CPAP. The study is instrumental in identifying the optimal OSA therapy for Veterans with PTSD and the OSA phenotype that would predict oral appliance response

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a prevalent disorder associated with poor neurocognitive performance and organ system dysfunction due to intermittent hypoxia and repeated arousals. The repetitive hemodynamic stresses are implicated in the increased incidence of systemic hypertension and cardiovascular diseases. Insufficient and disrupted sleep has similar negative impact on mood, attention, cognition, and behavior. In Veterans with post traumatic stress disorder (PTSD), the disturbed sleep can worsen further the cognitive-behavioral manifestations of PTSD and contributes to poor mental and physical health outcomes. Recent epidemiologic studies largely support the association of higher rates of OSA in patients with PTSD compared with the general population. Treatment of the underlying obstructive sleep disturbances with continuous positive airway pressure (CPAP) has resulted in restoration of sleep architecture, decrease daytime sleepiness, and reduction in nightmares frequency and intensity. However, adherence to treatment with CPAP is less than optimal in Veterans with PTSD. Mandibular advancing devices (MADs) are considered non surgical alternatives to CPAP and are preferred in a head to head comparison to CPAP in OSA subjects without PTSD. However, there has been no study to the investigators' knowledge that has assessed MAD in terms of clinical efficacy, compliance, and quality of sleep compared to CPAP in OSA patients with PTSD. Therefore, the investigators hypothesize that MAD is not inferior to CPAP in treating OSA effectively in Veterans with PTSD and OSA. To that end, the investigators propose to conduct a feasibility study using a randomized crossover trial of 12 weeks of CPAP and MAD in 42 consecutive outpatients with PTSD newly diagnosed with OSA separated by 2 weeks washout period.

The primary endpoint of the trial is to compare the treatment efficacy of CPAP and MAD in Veterans with PTSD and OSA. Secondary endpoints aim at: 1) comparing change in the Epworth Sleepiness Scale, SF-36, and the Pittsburgh Sleep Quality Index at end of treatment following use of CPAP versus MAD, 2) comparing adherence and short-term side effects between using CPAP and MAD in PTSD patients with OSA, and 3) determining anthropomorphic, polysomnographic, and cephalometric predictors of successful MDA response. Assessments at the end of both limbs comprise evaluation of quality of sleep, daytime sleepiness, quality of life, and side effects of treatment. Compliance with each therapy will be measured at the end of each treatment period.

The results of the trial are pivotal in determining the efficacy, tolerability, and adherence to MAD compared to CPAP in Veterans with PTSD and OSA. This feasibility study would form the basis of a future trial examining the effectiveness of various therapeutic modalities for OSA on PTSD symptomatology and progression.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients aged 18-70 years of age
* Documented obstructive sleep apnea by polysomnography (AHI 5 or more/hr)
* Established diagnosis of PTSD related to any past lifetime traumatic event and have a diagnosis of current, chronic PTSD

Exclusion Criteria:

* Central sleep apnea defined as central apnea/hypopnea >50% of the total respiratory events
* Prior treatment for sleep apnea
* Veterans with fewer than 4 teeth remaining in either arch
* Coexisting narcolepsy
* Tempo-mandibular joint disease
* Epilepsy
* Prominent suicidal or homicidal ideation
* Diagnosis of dementia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-11-01 (Actual); Primary Completion 2016-10-30 (Actual); Study Completion 2017-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ali A El-Solh, MD MPH, Principal Investigator — VA Western New York Healthcare System, Buffalo, NY
Locations (1):
- VA Western New York Healthcare System, Buffalo, NY, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El-Solh AA, Homish GG, Ditursi G, Lazarus J, Rao N, Adamo D, Kufel T. A Randomized Crossover Trial Evaluating Continuous Positive Airway Pressure Versus Mandibular Advancement Device on Health Outcomes in Veterans With Posttraumatic Stress Disorder. J Clin Sleep Med. 2017 Nov 15;13(11):1327-1335. doi: 10.5664/jcsm.6808. PMID 29065960

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 127 Veterans were considered for study participation between August 2013 and April 2016. Fifty-four patients agreed to enroll in the study but twelve patients either failed to return for scheduled visits or withdrew from further participation because of lack of time or other pressing matters. Forty-two were randomized to CPAP or MAD.
Period: First Intervention
Arm/Group | CPAP First, MAD | MAD First, CPAP
Started | 21 | 21
Completed | 19 | 20
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1
Period: Second Intervention
Arm/Group | CPAP First, MAD | MAD First, CPAP
Started | 19 | 20
Completed | 17 | 18
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants were asked to acclimate to CPAP and MAD for 4 weeks (total) during which adjustments to both modes of therapy are made aiming to optimize comfort and abolish snoring.
  If the interface was found to be uncomfortable, the patient was given the opportunity to change the mask. None of the participants was exposed to dual therapy or had access to both devices at the same time. Weekly phone calls were made to inquire about side effects or problems with CPAP or MAD. At the end of the acclimatization period, patients underwent a 2-week washout, after which they were randomly assigned in 1:1 ratio via a presealed and numbered opaque white envelope to one of the two treatment modalities (CPAP or MAD) that included the assignment to receive 12 weeks of treatment with MAD and CPAP in alternating order
Arm/Group | All Study Participants
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Residual Apnea Hypopnea Index
Description: The primary endpoint of the study was tested by comparing the upper limit of the 95% confidence interval for the CPAP-MAD difference in residual AHI with the a priori noninferiority margin using the paired t test
Time Frame: up to 12 weeks
Measure: Mean (Standard Deviation); unit: events per hour
Groups:
- CPAP: CPAP treatment for sleep apnea
  CPAP: CPAP Treatment for 12 weeks
- Mandibular Advancing Device: MAD treatment for sleep apnea
  MAD: MAD Treatment for 12 weeks
Arm/Group | CPAP | Mandibular Advancing Device
Number analyzed (Participants) | 35 | 35
events per hour | 3.9 (4.8) | 26.3 (25.6)
Statistical Analysis 1: Comparison: CPAP vs Mandibular Advancing Device; Test type: Equivalence — The primary endpoint of the study was tested by comparing difference in residual AHI using the paired t test; p < 0.001, t-test, 2 sided

2. Secondary Outcome: Health Outcomes
Description: Health outcomes including ESS, PCL-M, and PSQI. ESS is a short questionnaire validated to measure excessive daytime sleepiness in patients with OSA 17. It measures the likelihood of falling asleep in eight different situations, with a score of 0-3 for each situation. The sum of individual scores for the eight items gives the final ESS score, ranging from 0-21. An ESS score >10 suggests excessive daytime sleepiness (EDS). The PSQI is a self-rating questionnaire that consists of seven dimensions. The possible scores range from 0-21, with greater than five indicative of impaired sleep quality. The PTSD Checklist is a 17-item self-report measure (1-5 points each) that assesses PTSD symptoms in relation to stressful military experiences. PTSD symptom severity scores are determined by summing the participants' answers to all 17 items from 1 ("not at all") to 5 ("extremely")(range 17-85) 14 with 5-10 point change indicating statistically significant response to treatment
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Mandibular Advancing Device: Mandibular advancing device treatment for 12 weeks
Arm/Group | CPAP | Mandibular Advancing Device
Number analyzed (Participants) | 35 | 35
units on a scale
  Epworth Sleepiness Scale | 9.4 (4.7) | 9.5 (4.9)
  PTSD Checklist | 49.9 (15.4) | 50.03 (13.64)
  Pitt sleep quality index | 17.3 (0.2) | 17.3 (0.2)
Statistical Analysis 1: Comparison: CPAP vs Mandibular Advancing Device; ESS; Test type: Equivalence — t test assuming unequal variance; p = 0.97, t-test, 2 sided
Statistical Analysis 2: Comparison: CPAP vs Mandibular Advancing Device; PCL; Test type: Equivalence — t test assuming unequal variance; p = 0.98, t-test, 2 sided
Statistical Analysis 3: Comparison: CPAP vs Mandibular Advancing Device; PSQI; Test type: Equivalence — t-test assuming non unequal variance; p = 0.31, t-test, 2 sided

3. Secondary Outcome: General Health SF-36
Description: The SF-36 is a generic 36-item Short Form Medical Outcomes Survey (SF-36) 16. It has eight main domains: physical functioning, role limitation due to physical problems, role limitation due to emotional problems, social functioning, mental health, energy/vitality, bodily pain, and general health perception. General Health SF36 score is coded, summed, and transformed onto a scale from 0 to 100 (worst to best possible health).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CPAP | Mandibular Advancing Device
Number analyzed (Participants) | 35 | 35
units on a scale | 49.33 (17.09) | 50.58 (15.45)
Statistical Analysis 1: Comparison: CPAP vs Mandibular Advancing Device; Test type: Equivalence — t test assuming unequal variance; p = 0.54, t-test, 2 sided

4. Secondary Outcome: Adherence to Therapy
Description: comparison of the number of hours per night used while on CPAP versus MAD
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: hours per night
Arm/Group | CPAP | Mandibular Advancing Device
Number analyzed (Participants) | 35 | 35
hours per night | 3.4 (2.48) | 5.66 (2.43)
Statistical Analysis 1: Comparison: CPAP vs Mandibular Advancing Device; Test type: Equivalence — t test assuming unequal variance; p < 0.001, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | CPAP | Mandibular Advancing Device
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 26/35 | 14/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CPAP (N=35) | Mandibular Advancing Device (N=35)
mask discomfort (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 0 (0)
claustrophobia (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 0 (0)
Jaw pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 9 (9)
Dry mouth (General disorders) | 10 (10) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes